CLINICAL TRIAL: NCT01212432
Title: Daptomycin Pharmacokinetics in Critically Ill Patients Undergoing Continuous Veno-venous Hemodiafiltration, a Dose Finding Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Maggiorini Marco, Prof. Dr. med., University Hospital Zurich, Intensivmedizin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAPTO_CH08
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-07

CONDITIONS: Gram-Positive Bacterial Infections
Keywords: Gram positive infection and CRRT
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Daptomycin kinetics in CRRT

SUMMARY:
Daptomycin kinetics in CRRT

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* male or female of 18 years or older
* females: negative pregnancy test
* Hospitalisation in the medical ICU
* High suspicion or evidence of Gram-positive infections requiring antibiotic therapy
* Subjects receiving standard antibiotic treatment for Gram-positive infection
* Evidence of renal failure
* Clinical necessity for continuous renal replacement therapy
* Written informed consent signed by the patient or a next of kin and an independent physician in case the patient is not able to sign.

Exclusion criteria:

* Skeletal muscle disorders or CPK levels of > 2 x ULN
* History of hypersensitivity to the drug
* Participation in another study
* Subjects with a history of muscle disease
* Patients with severe liver function impairment (Child
* Life expectancy of less than 5 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics | 2011

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland